CLINICAL TRIAL: NCT04037930
Title: Changes in Cardiovascular Response and Dental Anxiety in Multiple Implant Surgery
Brief Title: Cardiovascular Response in Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, Principal investigator, Erzincan University
Other Study IDs: erzincan binali yıldırım ç
Record Dates: First submitted 2019-07-28; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Dental Anxiety; Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: multiple implant surgery — Patients older than 30 years who will undergo elective dental implant surgery.

SUMMARY:
The aim of this study was to observe the level of anxiety and its relationship with cardiovascular changes in each implant.

ELIGIBILITY:
Inclusion Criteria:

* Over 30
* 4 years and older implant in the same session

Exclusion Criteria:

* patients with syndrome,
* having systemic disease,
* having heart problems,
* undergo another oral or maxillofacial procedure in the last 6 months,
* using medications that may cause changes in medical conditions and heart rate,

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients over the age of 30 undergoing elective dental implant surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 4 months
  cardiovascular changes in implant surgery

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corah NL. Development of a dental anxiety scale. J Dent Res. 1969 Jul-Aug;48(4):596. doi: 10.1177/00220345690480041801. No abstract available. PMID 5256508
- [Result] CANDIDO, Milene Cardoso, et al. Clinical setting influences physiological responses in dental implant patients. Brazilian Journal of Oral Sciences, 2014, 13.2: 109-113.
- [Result] Newton JT, Buck DJ. Anxiety and pain measures in dentistry: a guide to their quality and application. J Am Dent Assoc. 2000 Oct;131(10):1449-57. doi: 10.14219/jada.archive.2000.0056. PMID 11042984
- [Result] Nagao H, Munakata M, Tachikawa N, Shiota M, Kasugai S. [Clinical study of risk management for dental implant treatment--changes of blood pressure and pulse rate during implant surgery under local anesthesia]. Kokubyo Gakkai Zasshi. 2002 Mar;69(1):27-33. doi: 10.5357/koubyou.69.27. Japanese. PMID 11968835